CLINICAL TRIAL: NCT04398342
Title: A Descriptive Study of Children With Cerebral Palsy Participating in The Danish Cerebral Palsy Follow-Up Program, With Emphasis on Their Hip Status
Brief Title: Characteristics of Children With Cerebral Palsy Who Develops Hip Displacement in Denmark
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mette Røn Kristensen (Other)
Responsible Party: Sponsor-Investigator, Mette Røn Kristensen, Regional coordinator for CPOP in the capital region of Denmark, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Other Study IDs: P-2019-143 1
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy; Hip Displacement; Hip Dislocation; Child; Registries; Orthopedic; Radiography
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Cerebral Palsy in Denmark: Children diagnosed with cerebral palsy born 2003 - 2020 and registered in the Danish Cerebral Palsy Follow-up Program.

SUMMARY:
The aim is to describe the characteristics of children with cerebral palsy in Denmark. Furthermore, we want to focus on status of the children's hips.

DETAILED DESCRIPTION:
Introduction: In 1994, a surveillance programme for children with Cerebral Palsy called the Cerebral Palsy Follow-Up Programme (CPUP) was established in Sweden with the primary purpose of preventing hip dislocation.

Hip dislocation is a serious complication to cerebral palsy, which is very painful for the child and requires complex hip surgery. Research studies have documented the effects of the follow-up program on the prevention of dislocation of the hip in children with CP in Sweden.

In 2003, the region of Southern Denmark introduced the Swedish follow-up program with the Danish name Cerebral Palsy Follow-up Program (CPOP). CPOP has since become a national follow-up program as well as a national clinical quality database in Denmark that includes children with CP aged 0-15 years and children with cerebral palsy-like symptoms aged 0-5 (5). The objective of the CPOP is to prevent complications associated with CP such as hip dislocation, scoliosis and contractures of muscles and joints.

It is now ten years since the first children were included in CPOP. There is no report describing the characteristics of children with cerebral palsy in Denmark and the status of the primary aim of the programme, hip status.

This study includes children diagnosed with CP born 2003 - 2020 and registered in the Danish Cerebral Palsy Follow-up Program.

Variables that will be analyzed are:

* age,
* Gross Motor Function Classification System Level I-V
* cerebral palsy subtype,
* Acetabular index,
* standing function,
* range of motion (hip abduction, hip extension, hip external rotation, hamstrings length)
* Modified Ashworth Scale (hip adduction, hip flexion, knee extension)
* Functional Mobility Scare (FMS)
* Gross Motor Function Measure (GMFM)
* hip displacement. Hip displacement is measured using divided into three categories; MP < 33 %, MP > 33-39 % og MP > 40 % with an extra category MP 100% describing children with hip dislocation.
* hip surgery. Categorized as; 1) soft tissue surgery, 2) neurosurgical procedures 3) osseous procedures.

Data will be obtained from the national clinical quality database the Danish Cerebral Palsy Follow-up Program and the Danish National Patient Register.

Variables will be summarize by counts, proportions and/or percentages using graphs and tables. Furthermore, the median and interquartile range will be specified when meaningful. Additionally, we will do non-parametric statistics (significance tests).

Currently, we do not have information about the extent of missing data for the different variables. When we have obtained the data, we will determine whether we have sufficient completeness for these variables to be included and reported in the statistical significance tests.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with CP born 2003 - 2020
* Classified at Gross Motor Function Classification Level I to V
* Minimum one radiographic examination of the hips.

Exclusion Criteria:

- Cerebral palsy diagnosis was not confirmed.

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children registered in the Danish Cerebral Palsy Follow-up Program.
Sampling Method: Non-Probability Sample
Enrollment: 957 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2020-12-27 (Estimated)

PRIMARY OUTCOMES:
Characteristics for children with CP in Denmark | Through study completion, on average 3 years
  Age, Gross Motor Function Classification Level (I-V), cerebral palsy subtype, acetabular index, standing function, Functional Mobility Scale, Gross Motor Function Measure, range of motion (hip abduction, hip extension, hip external rotation, hamstrings length), Modified Ashworth Scale (hip adduction, hip flexion, knee extension), hip displacement ( Migration Percentage) and hip surgery.

SECONDARY OUTCOMES:
Association between Gross Motor Function Classification System and Migrations Percentage (MP) | Through study completion, on average 3 years
  Gross Motor Function Classification System and Migration Percentage
Association between cerebral palsy subtype and Migrations Percentage | Through study completion, on average 3 years
  cerebral palsy subtype and Migrations Percentage
Association between standing position and Migrations Percentage | Through study completion, on average 3 years
  Variables for standing position and Migrations Percentage
Association between range of motion and Migrations Percentage | Through study completion, on average 3 years
  range of motion (hip abduction, hip extension, hip external rotation, hamstrings length) and Migrations Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Mette Røn Kristensen, PT, MSc, Principal Investigator — Fysio- og Ergoterapien, afsnit 234-236, Hvidovre Hospital,
Locations (1):
- Fysio- og Ergoterapien, afsnit 234-236, Hvidovre hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen HM, Nordbye-Nielsen K, Moller-Madsen B, Johansen M, Ellitsgaard N, Pedersen CR, Rackauskaite G, Engberg H, Pedersen NW. The Danish Cerebral Palsy Follow-up Program. Clin Epidemiol. 2016 Oct 25;8:457-460. doi: 10.2147/CLEP.S99474. eCollection 2016. PMID 27822084
- [Background] Hagglund G, Alriksson-Schmidt A, Lauge-Pedersen H, Rodby-Bousquet E, Wagner P, Westbom L. Prevention of dislocation of the hip in children with cerebral palsy: 20-year results of a population-based prevention programme. Bone Joint J. 2014 Nov;96-B(11):1546-52. doi: 10.1302/0301-620X.96B11.34385. PMID 25371472